CLINICAL TRIAL: NCT01063322
Title: New Techniques to Evaluate Mitral Regurgitation
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100039; 10-H-0039
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2018-04-11

CONDITIONS: Mitral Valve Regurgitation
Keywords: Mitral Regurgitation; Echocardiography; Cardiac Magnetic Resonance; Regurgitant Volume; Mitral Valve Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Mitral regurgitation, or leaking of the mitral heart valve, is usually studied and assessed with an ultrasound test called a two-dimensional (2D) echocardiogram. While this test has proved very useful, technological improvements have helped researchers develop ways to study the heart valves using imaging with three-dimensional (3D) capabilities. In addition, recently developed magnetic resonance imaging (MRI) techniques may be able to provide better information about the causes and severity of the leak. Researchers are interested in testing these new techniques to determine their usefulness for patients with mitral regurgitation.

Objectives:

- To evaluate newer methods of studying mitral regurgitation severity using real-time 3D echocardiography (RT3DE) and cardiac magnetic resonance imaging (CMRI).

Eligibility:

- Individuals at least 21 years of age who have been diagnosed with more than mild mitral regurgitation.

Design:

* Participants will have two procedures as part of this study: an echocardiogram and an MRI scan.
* For the echocardiogram, participants will have an ultrasound scan with a special kind of probe. Participants may also receive an injection of a contrast agent to provide a better image of the heart on the scan. The scan will take approximately 1 hour to complete.
* For the MRI scan, participants will have a standard MRI with special pads placed on the chest to provide better imaging of the heart. The scan will usually take between 45 and 90 minutes to complete.

DETAILED DESCRIPTION:
Echocardiography is currently the technique of choice to assess the etiology and severity of mitral regurgitation (MR). Multiple 2D and Doppler parameters are assessed in an integrated fashion and the proximal flow convergent zone of the mitral regurgitation jet is used to calculate effective regurgitant orifice area and regurgitant volume. These measurements have been shown to have important prognostic information. In the last two years, the development of transesophageal imaging with 3D capability has allowed a better visualization of mitral leaflet pathology. Color Doppler 3D studies have shown that 2D methods generally underestimate mitral regurgitant volume. Magnetic resonance techniques have recently been developed to quantitate flow and calculate regurgitant volumes.

The purpose of this study is to evaluate newer methods of quantitating mitral regurgitation severity using real-time 3D echocardiography (RT3DE) and cardiac magnetic resonance imaging (CMR). Although RT3DE measurements have been shown to correlate well with CMR measures of LV volumes, using a 3D volumetric method to calculate mitral regurgitant volumes has not been well studied. In patients with more than mild mitral regurgitation, we will obtain transthoracic RT3DE measures of mitral regurgitant volume and compare them with traditional 2D measures of MR severity. We will also compare RT3DE and CMR measures of mitral regurgitant volume.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult patient, age greater than or equal to 21 years
* Able to give written informed consent
* Prior cardiac testing clinically read as having greater than mild MR

EXCLUSION CRITERIA:

* Atrial fibrillation or other irregular rhythm that would preclude adequate 3D image acquisition
* History of valve surgery or significant valve disease other than mitral regurgitation
* Patients with pacemakers, defibrillators, cerebral aneurysm clips, neural stimulators, ear implants or other clinical contra-indications for magnetic resonance scanning will be excluded from the CMR portion of the study
* Any unstable condition that would make additional imaging time inadvisable (in the opinion of the investigator or managing physician)
* Pregnant or lactating women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-02-01; Study Completion 2018-04-11

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Sachdev, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Sheikh K, Smith SW, von Ramm O, Kisslo J. Real-time, three-dimensional echocardiography: feasibility and initial use. Echocardiography. 1991 Jan;8(1):119-25. doi: 10.1111/j.1540-8175.1991.tb01409.x. PMID 10149247
- [Background] Schmidt MA, Ohazama CJ, Agyeman KO, Freidlin RZ, Jones M, Laurienzo JM, Brenneman CL, Arai AE, von Ramm OT, Panza JA. Real-time three-dimensional echocardiography for measurement of left ventricular volumes. Am J Cardiol. 1999 Dec 15;84(12):1434-9. doi: 10.1016/s0002-9149(99)00591-3. PMID 10606118
- [Background] Jacobs LD, Salgo IS, Goonewardena S, Weinert L, Coon P, Bardo D, Gerard O, Allain P, Zamorano JL, de Isla LP, Mor-Avi V, Lang RM. Rapid online quantification of left ventricular volume from real-time three-dimensional echocardiographic data. Eur Heart J. 2006 Feb;27(4):460-8. doi: 10.1093/eurheartj/ehi666. Epub 2005 Nov 30. PMID 16319085